CLINICAL TRIAL: NCT03079518
Title: Intravenous Iron in paTients With Heart failURe and Reduced Ejection fracTion (HFREF) pLus Iron dEficiency: Effects Upon Phosphate and FGF23 Metabolism
Brief Title: Intravenous Iron in paTients With Heart failURe and Reduced Ejection fracTion (HFREF) pLus Iron dEficiency
Acronym: Iron Turtle
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: RWTH Aachen University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 16-047
Record Dates: First submitted 2017-03-03; First posted 2017-03-14 (Actual); Last update posted 2017-12-06 (Actual); Status verified 2017-12

CONDITIONS: Heart Failure, Systolic; Iron Deficiency
Keywords: iron deficiency; HFREF; FGF23; ferric carboxymaltose
MeSH Terms: conditions — Heart Failure, Systolic; Iron Deficiencies | interventions — ferric carboxymaltose

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patients with HFREF & CKD (Active Comparator): treated with intravenous single-shot 1000mg Ferric Carboxymaltose infusion; additional intervention: blood withdrawal
  Interventions: Drug: Ferric Carboxymaltose; Other: blood withdrawal
- Patients with HFREF (Active Comparator): treated with intravenous single-shot 1000mg Ferric Carboxymaltose infusion; additional intervention: blood withdrawal
  Interventions: Drug: Ferric Carboxymaltose; Other: blood withdrawal

INTERVENTIONS:
Drug: Ferric Carboxymaltose — single shot infusion
  Other Names: Ferinject
Other: blood withdrawal — for determination of serum and urinary biomarkers of chronic kidney disease metabolism and other parameters

SUMMARY:
Effects of ferric carboxymaltose single HD (1000 mg) infusion upon FGF23 in patients with isolated HFREF compared to patients with HFREF+CKD (all pts with iron deficiency). This study aims at identification of the optimal target population for a follow-up ("main") study.

DETAILED DESCRIPTION:
Iron deficiency is highly prevalent in patients with HFREF and intravenous high-dose (HD) iron application has significantly improved clinically meaningful endpoints in such patients. The best evidence is existent for ferric carboxymaltose. Intravenous HD iron may influence phosphate metabolism via increases in levels of intact FGF23 and hence induce prolonged hypophosphatemia. Such increases in FGF23 may particularly occur depending on the type of iron carrier.

FGF23 is a significant risk factor for mortality and morbidity in patients with HFREF and other cardiac populations at risk and may directly cause left ventricular hypertrophy and dysfunction. Hence, the application of i.v. HD iron may have potentially beneficial effects on cardiac function but harmful effects via FGF23-induction and hypophosphatemia at the same time. However, FGF23 metabolism has not yet been evaluated in HFREF patients following i.v. HD iron.

FGF23 is elevated in patients with chronic kidney disease. Patients with HFREF + CKD = chronic cardio-renal syndrome are at particular risk regarding elevated morbidity and mortality. The effects of intravenous HD iron upon phosphate and FGF23 metabolism in patients with HFREF + CKD is unknown and effects in this setting may be different compared to effects in patients without pre-existing FGF23 stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent.
* Age > 18 yrs
* Symptomatic HFREF (LV ejection fraction < 45%) with optimal medical therapy (OMT) for at least 2 months
* Iron deficiency as indicated by by ferritin <100 ng/mL or ferritin 100-299 ng/ml when transferrin saturation (TSAT) <20% and Hb value < 13mg/dl (women) and <14 mg/dl (men)
* Group A: Stable CKD for at least 2 months, defined by estimated glomerular filtration rate (eGFR) (CKD-EPI formula) as 15-60 ml/min/1,73 m3 (CKD III, IV, V-non D)
* Group B: patients with stable eGFR > 60 ml/min/1,73 m3

Exclusion Criteria:

* Known hypersensitivity to ferric carboxymaltose or any constituents of the formulation,
* Plasma Phosphate < 2.5 mg/dL at screening,
* Renal replacement therapy/transplantation,
* Pregnancy or lactation
* iron substitution therapy or erythropoetin (epo) therapy within 6 weeks before
* participation in another clinical trial with an experimental drug
* expectation of missing compliance
* alcohol or drug abuse
* The subject is mentally or legally incapacitated
* patients who are in a relationship of dependence or in a working relationship to the sponsor, the investigator or his representative

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2017-03-10 (Actual); Primary Completion 2017-10-25 (Actual); Study Completion 2017-10-25 (Actual)

PRIMARY OUTCOMES:
changes in blood intact FGF23 after infusion of 1000 mg ferric carboxymaltose | 4 weeks
  intact FGF23 concentration in kRU/l
changes in blood c-term FGF23 after infusion of 1000 mg ferric carboxymaltose | 4 weeks
  c-terminal FGF23 concentration in kRU/l

SECONDARY OUTCOMES:
changes of serum biomarkers of chronic kidney disease metabolism | 4 weeks
  PTH, Vitamin D, ALP, s-klotho, PINP, proBNP
changes of urinary marker of tubular damage | 4 weeks
  NGAL, KIM-1
phosphate level | 4 weeks
  < 1,25 mg/dL
changes of Inflammatory mediators | 4 weeks
  IL1, IL6, TNF-alpha, hsCRP

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Medicine, Division of Cardiology, Pulmonary Diseases and Vascular Medicine at the University Hospital, RWTH Aachen, Aachen, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared due to publication afterwards

REFERENCES:
- [Derived] Stohr R, Sandstede L, Heine GH, Marx N, Brandenburg V. High-Dose Ferric Carboxymaltose in Patients With HFrEF Induces Significant Hypophosphatemia. J Am Coll Cardiol. 2018 May 15;71(19):2270-2271. doi: 10.1016/j.jacc.2018.03.448. No abstract available. PMID 29747838